CLINICAL TRIAL: NCT00968513
Title: Evaluation of Tobacco Treatment Strategies for Inpatient Psychiatry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Prochaska, Associate Professor in Residence, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH083684 (NIH); R01MH083684 (NIH); DAHBR A2-AID (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation, Inpatient Psychiatry, Stages of Change
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: NRT
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (Active Comparator): (N=132) brief cessation advice, a quit smoking guide, and nicotine replacement provided during hospitalization
  Interventions: Behavioral: Usual Care
- Brief Treatment (Experimental): (N=416) adds a stage-based manual, computer-delivered stage-tailored individualized feedback and brief cessation counseling sessions during hospitalization and repeated at months 3 and 6, and access to 12 weeks of nicotine replacement following hospitalization.
  Interventions: Behavioral: Brief Intervention
- Extended Treatment (Experimental): (N=408) builds upon our current brief treatment and provides 12 additional weeks of nicotine replacement (24 weeks total) with individualized, counselor-delivered motivational and manualized cognitive behavioral cessation treatment.
  Interventions: Behavioral: Extended Treatment

INTERVENTIONS:
Behavioral: Brief Intervention — (N=416) adds a stage-based manual, computer-delivered stage-tailored individualized feedback and brief cessation counseling sessions during hospitalization and repeated at months 3 and 6, and access to 12 weeks of nicotine replacement following hospitalization
  Arms: Brief Treatment
Behavioral: Extended Treatment — (N=408) builds upon our current brief treatment and provides 12 additional weeks of nicotine replacement (24 weeks total) with individualized, counselor-delivered motivational and manualized cognitive behavioral cessation treatment.
  Arms: Extended Treatment
Behavioral: Usual Care — (N=132) brief cessation advice, a quit smoking guide, and nicotine replacement provided during hospitalization
  Arms: Usual Care

SUMMARY:
This study aims to evaluate, in a randomized controlled trial, tobacco treatments of varying intensities for smokers hospitalized on acute psychiatric inpatient units.

DETAILED DESCRIPTION:
Using a three group additive design, this randomized clinical trial (N=956) aims to evaluate tobacco cessation treatments of varying intensities initiated in the acute psychiatric inpatient setting. The three groups are:

1. Usual Care (N=132) consisting of brief cessation advice, a quit smoking guide, and nicotine replacement provided during hospitalization;
2. Brief Treatment (N=416) adds a stage-based manual, computer-delivered stage-tailored individualized feedback and brief cessation counseling sessions during hospitalization and repeated at months 3 and 6, and access to 12 weeks of nicotine replacement following hospitalization;
3. Extended Treatment (N=408) builds upon our current brief treatment and provides 12 additional weeks of nicotine replacement (24 weeks total) with individualized, counselor-delivered motivational and manualized cognitive behavioral cessation treatment.

This study seeks to determine: (i) whether the initial successes seen in an academic-based psychiatric hospital can be replicated in a larger and more diverse patient population; and (ii) if more extended and intensive treatment combining nicotine replacement therapy (NRT) with individualized, counselor-delivered motivational and manualized cessation-focused cognitive behavioral counseling (CBT) can outperform our current best practices. Ultimately, this research could lead to a model smoking cessation intervention for smokers with severe mental illness and, more generally, may provide a useful model for understanding the nature and complexity of intervening on comorbidities.

We hypothesize that the extended treatment will outperform the brief treatment, and that both treatment groups will be more effective than usual care in producing quit attempts and ultimately abstinence from cigarettes. Secondary specific aims will model the cost-effectiveness and budgetary impacts of the treatment conditions; examine moderators and mediators of treatment outcomes; and prospectively examine the relation between changes in smoking, mental health functioning, and use of other substances over time.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be men and women 18 years of age and older, recruited from four acute inpatient psychiatry units at the Alta Bates Summit Medical Center - Herrick Campus, located in Berkeley, CA, one acute inpatient psychiatry unit at Langley Porter Psychiatric Institute, located in San Francisco, CA, and two acute inpatient psychiatry units at Stanford Hospital, located in Stanford, CA. Inclusion criteria are: smoking 5 or more cigarettes per day and at least 100 cigarettes in one's lifetime, no plan to relocate outside of the greater Bay Area in the next 18 months, and telephone access for scheduling follow-up assessments.

Exclusion Criteria:

* Study exclusion criteria are: dementia or other brain injury precluding ability to participate; non-English speaking; complete homelessness; pregnancy or breastfeeding, and active ulcer disease (PUD). The relationship between nicotine and ulcers is a theoretical concern and our approach to now exclude patients with active ulcer disease is conservative. There is no data to show NRT causes/worsens ulcers. Recruitment of acutely psychotic, manic, or hostile patients will be delayed until there is significant reduction of these symptoms and patients are able to consent to study participation. Threats of violence in particular are taken seriously, and patients will not be recruited if they may be a threat to study staff in the outpatient setting. At this point, non-English measurement and intervention materials are not available. Pregnant smokers will be referred out for more specialized behavioral treatments. Exclusionary criteria are purposefully minimal in order to maximize information about treating tobacco dependence in smokers in inpatient psychiatry. The study sample is anticipated to be diverse with respect to gender and ethnicity, educational and socioeconomic level, and psychiatric diagnoses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 956 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith J. Prochaska, PhD, MPH, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Alta Bates Summit Medical Center, Berkeley, California
  - UCSF Langley Porter Psychiatric Institute, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prochaska JJ, Grana RA. E-cigarette use among smokers with serious mental illness. PLoS One. 2014 Nov 24;9(11):e113013. doi: 10.1371/journal.pone.0113013. eCollection 2014. PMID 25419703
- [Derived] Schuck RK, Dahl A, Hall SM, Delucchi K, Fromont SC, Hall SE, Bonas T, Prochaska JJ. Smokers with serious mental illness and requests for nicotine replacement therapy post-hospitalisation. Tob Control. 2016 Jan;25(1):27-32. doi: 10.1136/tobaccocontrol-2014-051712. Epub 2014 Sep 10. PMID 25209524
- [Derived] Prochaska JJ, Fromont SC, Delucchi K, Young-Wolff KC, Benowitz NL, Hall S, Bonas T, Hall SM. Multiple risk-behavior profiles of smokers with serious mental illness and motivation for change. Health Psychol. 2014 Dec;33(12):1518-29. doi: 10.1037/a0035164. Epub 2014 Jan 27. PMID 24467257

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual Care: brief cessation advice, a quit smoking guide, and nicotine replacement provided during hospitalization
- Brief Treatment: Brief Intervention: adds a stage-based manual, computer-delivered stage-tailored individualized feedback and brief cessation counseling sessions during hospitalization and repeated at months 3 and 6, and access to 12 weeks of nicotine replacement following hospitalization
- Extended Treatment: Extended Treatment: builds upon our current brief treatment and provides 12 additional weeks of nicotine replacement (24 weeks total) with individualized, counselor-delivered motivational and manualized cognitive behavioral cessation treatment.
Period: Overall Study
Arm/Group | Usual Care | Brief Treatment | Extended Treatment
Started | 132 | 416 | 408
Completed | 128 | 406 | 393
Not Completed | 4 | 10 | 15
Not completed — Death | 4 | 10 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Brief Treatment | Extended Treatment | Total
Number analyzed (Participants) | 132 | 416 | 408 | 956
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 130 | 404 | 397 | 931
  >=65 years | 2 | 12 | 11 | 25
Age, Continuous [Mean (Full Range); unit: years] | 38 [18 to 68] | 39 [18 to 73] | 38 [18 to 71] | 39 [18 to 73]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 63 | 202 | 194 | 459
  Male | 67 | 209 | 211 | 487
  Transgender | 2 | 5 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 132 | 416 | 408 | 956

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Quit Smoking at 3, 6, 12, and 18 Months
Description: Number of Participants who Quit Smoking at 3, 6, 12, and 18 Months
Time Frame: 3, 6, 12, and 18 Month Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Brief Treatment | Extended Treatment
Number analyzed (Participants) | 132 | 416 | 408
Participants
  3 month | 13 | 70 | 63
  6 month | 15 | 75 | 78
  12 month | 21 | 78 | 74
  18 month | 17 | 80 | 82

2. Primary Outcome: Commitment to Abstinence
Description: Changes from one assessment point to the next in a Likert scale (1 to 10) measure of desire to quit smoking. 10 = strongest desire to quit.
Time Frame: baseline, 3, 6, 12, and 18 months
Population: Missing values at each timepoint per group were excluded from analyses.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Care | Brief Treatment | Extended Treatment
Number analyzed (Participants) | 132 | 416 | 408
score on a scale
  Baseline: number analyzed (Participants) | 132 | 415 | 408
  Baseline | 5.83 [1 to 10] | 6.20 [1 to 10] | 5.85 [1 to 10]
  3 month: number analyzed (Participants) | 82 | 257 | 254
  3 month | 6.27 [1 to 10] | 7.44 [1 to 10] | 7.09 [1 to 10]
  6 month: number analyzed (Participants) | 78 | 249 | 237
  6 month | 6.65 [1 to 10] | 7.22 [1 to 10] | 7.21 [1 to 10]
  12 month: number analyzed (Participants) | 78 | 227 | 229
  12 month | 7.06 [1 to 10] | 7.44 [1 to 10] | 7.33 [1 to 10]
  18 month: number analyzed (Participants) | 76 | 255 | 233
  18 month | 7.05 [1 to 10] | 7.47 [1 to 10] | 7.37 [1 to 10]

3. Primary Outcome: Number of Participants With Quit Attempts Lasting 24 Hours or More
Description: Number of participants with quit attempts lasting 24 hours or more at each follow up timepoint.
Time Frame: 3, 6, 12, and 18 months follow-up
Measure: Number; unit: participants
Groups:
- Brief Treatment: Brief Treatment: adds a stage-based manual, computer-delivered stage-tailored individualized feedback and brief cessation counseling sessions during hospitalization and repeated at months 3 and 6, and access to 12 weeks of nicotine replacement following hospitalization.
Arm/Group | Usual Care | Brief Treatment | Extended Treatment
Number analyzed (Participants) | 132 | 416 | 408
participants
  3 month | 42 | 181 | 162
  6 month | 40 | 169 | 149
  12 month | 47 | 156 | 170
  18 month | 47 | 183 | 165

ADVERSE EVENTS:
Time Frame: 18 months
Description: Participants assessed at 3, 6, 12 and 18 months for any AEs related to NRT use and for SAEs of hospitalization or ER presentation. Information on deaths were collected from family/friends/providers/etc.
Arm/Group | Usual Care | Brief Treatment | Extended Treatment
Serious Adverse Events (participants affected / at risk) | 105/132 | 308/416 | 310/408
Other Adverse Events (participants affected / at risk) | 17/132 | 120/416 | 126/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=132) | Brief Treatment (N=416) | Extended Treatment (N=408)
Placed on a 5150 (Psychiatric disorders) | 22 | 76 | 73
Placed on a 5250 (Psychiatric disorders) | 0 | 1 | 0
Accused of assault (Social circumstances) | 0 | 0 | 1
Ankle pain/injuries (Injury, poisoning and procedural complications) | 0 | 6 | 4
Ankle infection (Infections and infestations) | 1 | 0 | 0
Arm pain/injuries (Injury, poisoning and procedural complications) | 1 | 7 | 5
Arm infection (Infections and infestations) | 1 | 0 | 0
Injuries and treatment from assault excluding sexual assault (Injury, poisoning and procedural complications) | 2 | 7 | 6
Autoimmune disease (Immune system disorders) | 1 | 2 | 0
AWOL and re-admission (Social circumstances) | 0 | 1 | 0
Back pain/discomfort/injury (Injury, poisoning and procedural complications) | 3 | 10 | 8
Blood clot (Blood and lymphatic system disorders) | 1 | 1 | 2
Blood transfusion (Surgical and medical procedures) | 0 | 1 | 0
Bloodwork (Surgical and medical procedures) | 1 | 0 | 0
Hemoptysis (General disorders) | 0 | 0 | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1 | 3 | 1
Hypertension (Blood and lymphatic system disorders) | 1 | 2 | 2
Hypoglycemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypotension (Blood and lymphatic system disorders) | 0 | 1 | 2
Stroke (Blood and lymphatic system disorders) | 0 | 4 | 0
Brought into hospital by police (Social circumstances) | 0 | 3 | 1
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Congestive heart failure (Cardiac disorders) | 1 | 0 | 1
Heart attack (Cardiac disorders) | 0 | 0 | 2
Heart disease (Cardiac disorders) | 0 | 0 | 1
Heart pain (Cardiac disorders) | 0 | 2 | 1
Heart palpitations (Cardiac disorders) | 1 | 1 | 3
Cellulitis (Infections and infestations) | 1 | 1 | 1
Skin conditions (Skin and subcutaneous tissue disorders) | 3 | 1 | 5
Diagnostic (Surgical and medical procedures) | 2 | 3 | 2
Domestic violence (Social circumstances) | 1 | 2 | 1
Ear pain or other issues (Ear and labyrinth disorders) | 0 | 2 | 2
Ear infection (Infections and infestations) | 1 | 0 | 0
Eye pain or other issues (Eye disorders) | 2 | 0 | 5
Conjunctivitis (Infections and infestations) | 0 | 1 | 2
Face drooping and numb (General disorders) | 0 | 0 | 1
Facial pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Fall injury (Injury, poisoning and procedural complications) | 5 | 8 | 6
Foot pain/injury (Injury, poisoning and procedural complications) | 4 | 6 | 10
Foot infection (Infections and infestations) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Burst gallbladder (Hepatobiliary disorders) | 1 | 0 | 0
Constipation and bowel issues (Gastrointestinal disorders) | 2 | 2 | 3
Esophageal tear (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 4 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gential issues/pain (Reproductive system and breast disorders) | 2 | 3 | 6
Gential infection (Infections and infestations) | 0 | 0 | 1
Hand pain/injuries (Injury, poisoning and procedural complications) | 1 | 5 | 6
Hip pain/injuries (Injury, poisoning and procedural complications) | 1 | 3 | 0
Food and shelter (Social circumstances) | 1 | 4 | 9
Infected hair follicle (Infections and infestations) | 0 | 1 | 0
Unspecified infection (Infections and infestations) | 0 | 0 | 1
MRSA (Infections and infestations) | 0 | 0 | 1
Perirectal infection (Infections and infestations) | 0 | 1 | 0
Physical illness (Infections and infestations) | 0 | 1 | 0
Respiratory infection (Infections and infestations) | 1 | 2 | 5
Staph infection (Infections and infestations) | 0 | 0 | 2
Strep throat (Infections and infestations) | 0 | 1 | 1
Parasites (Infections and infestations) | 1 | 0 | 0
Insect bites (Infections and infestations) | 1 | 3 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Kidney issues (Renal and urinary disorders) | 0 | 2 | 3
Kidney infection (Infections and infestations) | 0 | 0 | 2
Leg pain/injuries (Injury, poisoning and procedural complications) | 4 | 7 | 12
Hospitalization in relation to legal issues (Social circumstances) | 1 | 2 | 0
Malaise (General disorders) | 2 | 4 | 2
IUD issues (Product Issues) | 0 | 1 | 0
pain at site of medical device (Product Issues) | 0 | 0 | 1
Medication complications (Product Issues) | 0 | 7 | 6
Medication management (Product Issues) | 1 | 2 | 5
Medication noncompliance (Social circumstances) | 10 | 34 | 31
Medication prescription (Social circumstances) | 0 | 7 | 2
Medication refill (Social circumstances) | 10 | 19 | 11
Mouth abscess or blister (Infections and infestations) | 1 | 1 | 0
Dystonia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pulled muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain/injuries (Injury, poisoning and procedural complications) | 0 | 3 | 2
Numbness in arm/leg (Nervous system disorders) | 0 | 2 | 1
Occupational injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Unsafe living conditions (Social circumstances) | 0 | 1 | 0
Having a strange sensation (General disorders) | 1 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1
Syncope (General disorders) | 3 | 5 | 3
Bladder infection (Infections and infestations) | 1 | 1 | 2
Bleeding stoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bowel blockage (Gastrointestinal disorders) | 1 | 0 | 0
Blood in urine/stool (Renal and urinary disorders) | 1 | 0 | 1
Blunt force trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Body aches (General disorders) | 0 | 1 | 0
Hemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cat scratches (Injury, poisoning and procedural complications) | 0 | 1 | 0
Chemical burn (Social circumstances) | 0 | 1 | 0
Chlamydia (Infections and infestations) | 0 | 1 | 0
Chronic conditions (General disorders) | 1 | 8 | 5
Colon inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Congestive heart failure (Cardiac disorders) | 0 | 0 | 1
Cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 6
Depression resulting from physical pain/condition (Psychiatric disorders) | 0 | 1 | 1
Diabetes (Metabolism and nutrition disorders) | 0 | 1 | 2
Diarhhea (Renal and urinary disorders) | 1 | 5 | 5
Dizziness (General disorders) | 2 | 1 | 3
Dog bite (Injury, poisoning and procedural complications) | 0 | 0 | 2
Edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Feeling unbalanced (General disorders) | 0 | 1 | 0
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Gallstones (Gastrointestinal disorders) | 0 | 1 | 0
Gangrene (Blood and lymphatic system disorders) | 0 | 0 | 1
Gonorrhea (Infections and infestations) | 0 | 1 | 0
Grave disability (General disorders) | 0 | 3 | 6
Head injury (Injury, poisoning and procedural complications) | 1 | 7 | 1
Headache (Nervous system disorders) | 1 | 7 | 6
Hepatitis C (Infections and infestations) | 0 | 1 | 0
Hernia (Gastrointestinal disorders) | 1 | 3 | 2
Liver issues (Hepatobiliary disorders) | 2 | 2 | 1
Loss of appetite (General disorders) | 0 | 1 | 0
Low oxygen level (Blood and lymphatic system disorders) | 0 | 0 | 1
Low potassium (Metabolism and nutrition disorders) | 0 | 3 | 0
Low sodium (Metabolism and nutrition disorders) | 0 | 1 | 0
Lower spine infection (Infections and infestations) | 0 | 0 | 1
Migraines (Nervous system disorders) | 1 | 4 | 6
MRI (Surgical and medical procedures) | 0 | 0 | 1
Mumps (Infections and infestations) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle tightness and weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nausea (General disorders) | 3 | 4 | 5
Neurothrombosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 1
Pinched nerve (Nervous system disorders) | 0 | 2 | 0
Poison ivy (Immune system disorders) | 0 | 0 | 1
Potassium deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0 | 0
Rectal bleeding (Injury, poisoning and procedural complications) | 0 | 1 | 1
Salt and electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Scabies (Infections and infestations) | 1 | 0 | 1
Sciatica (Injury, poisoning and procedural complications) | 1 | 1 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0
Shingles (Infections and infestations) | 0 | 0 | 1
Sore throat (General disorders) | 1 | 0 | 0
Sexually Transmitted Disease (Infections and infestations) | 0 | 1 | 1
Stitches/Sutures (Surgical and medical procedures) | 0 | 5 | 0
Sunburn (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Surgery (Surgical and medical procedures) | 3 | 12 | 4
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ulcer (General disorders) | 0 | 0 | 1
Unconscious in a public transportation station (Social circumstances) | 0 | 1 | 0
Uncontrollable nosebleed (General disorders) | 0 | 1 | 0
Weight loss (General disorders) | 0 | 0 | 1
Urinary issues/pain (Renal and urinary disorders) | 3 | 7 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 2
Vomiting (General disorders) | 1 | 6 | 7
Vomiting blood (General disorders) | 1 | 0 | 3
Abdominal pain/discomfort (Injury, poisoning and procedural complications) | 2 | 21 | 11
Arthritis pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chest pain/discomfort (Injury, poisoning and procedural complications) | 6 | 8 | 22
Dental pain (Injury, poisoning and procedural complications) | 1 | 7 | 2
Extreme pain in extremities (General disorders) | 0 | 0 | 1
Groin/Inguinal pain (Renal and urinary disorders) | 0 | 0 | 1
Hemorrhoid pain (Renal and urinary disorders) | 0 | 0 | 1
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Pain (unspecified) (General disorders) | 1 | 0 | 0
Pain due to neuropathy (Nervous system disorders) | 0 | 0 | 1
Pain from extreme cold (Social circumstances) | 0 | 1 | 0
Pain in hip joints (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in sides (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pain management (Surgical and medical procedures) | 0 | 0 | 1
Pelvis pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Physical pain (General disorders) | 1 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 4 | 1
Instant-onset dementia (Psychiatric disorders) | 1 | 0 | 0
Pain (Psychiatric disorders) | 0 | 1 | 0
Accused of hostile behavior (Social circumstances) | 0 | 1 | 0
Aggressive/hostile thoughts or behaviors (Psychiatric disorders) | 6 | 17 | 17
Agitation (Psychiatric disorders) | 1 | 9 | 7
Agoraphobia (Psychiatric disorders) | 0 | 0 | 1
Altered mental status (Psychiatric disorders) | 0 | 3 | 1
Anger/upset (Psychiatric disorders) | 2 | 5 | 6
Anxiety/nervousness (Psychiatric disorders) | 6 | 27 | 22
Behavior change and issues (Psychiatric disorders) | 4 | 12 | 16
Bipolar Disorder and related symptoms (Psychiatric disorders) | 1 | 3 | 1
Borderline Personality Disorder (Psychiatric disorders) | 0 | 1 | 0
Catatonia (Psychiatric disorders) | 0 | 0 | 1
Chest pain (Psychiatric disorders) | 0 | 3 | 1
Danger to self (Psychiatric disorders) | 2 | 14 | 13
Decreased motivation (Psychiatric disorders) | 0 | 0 | 1
Dehydration (Psychiatric disorders) | 0 | 0 | 1
Delusional thoughts/behaviors (Psychiatric disorders) | 3 | 10 | 7
Depression, saddness, grief (Psychiatric disorders) | 26 | 99 | 113
Destructive behavior (Psychiatric disorders) | 1 | 0 | 0
Disorganization, confusion (Psychiatric disorders) | 4 | 5 | 6
Dissociative episode (Psychiatric disorders) | 0 | 1 | 0
Eating disorder symptoms (Psychiatric disorders) | 1 | 3 | 4
Emotional distress, instability, problems (Psychiatric disorders) | 0 | 6 | 4
Feeling mentally unstable (Psychiatric disorders) | 0 | 1 | 0
Feeling unsafe (excluding domestic abuse) (Psychiatric disorders) | 0 | 4 | 5
Hallucinations (Psychiatric disorders) | 23 | 44 | 59
Homicidal ideation (Psychiatric disorders) | 6 | 16 | 16
Hysteria, grandiosity (Psychiatric disorders) | 0 | 1 | 0
Ideas of reference (Psychiatric disorders) | 1 | 0 | 0
Lack of self care (Psychiatric disorders) | 2 | 3 | 0
Malingering (Psychiatric disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 4 | 7 | 12
Mood swings; moodiness; worsening mood (Psychiatric disorders) | 2 | 0 | 3
Nervous/mental breakdown; Needing psychiatric care/observation (Psychiatric disorders) | 1 | 7 | 8
Out of body experience (Psychiatric disorders) | 1 | 0 | 0
Panic Attack (Psychiatric disorders) | 3 | 9 | 6
Paranoia (Psychiatric disorders) | 12 | 14 | 27
Psychiatric evaluation (Surgical and medical procedures) | 0 | 1 | 3
Psychosis/Psychotic behavior (Psychiatric disorders) | 6 | 11 | 13
PTSD (Psychiatric disorders) | 0 | 4 | 1
Racing thoughts (Psychiatric disorders) | 0 | 0 | 1
Rumination (Psychiatric disorders) | 0 | 0 | 1
Schizoaffective disorder; Shizophrenia symptoms (Psychiatric disorders) | 1 | 7 | 0
Stress (Psychiatric disorders) | 0 | 3 | 1
Substance use (Psychiatric disorders) | 23 | 48 | 50
Suicidal ideation (Psychiatric disorders) | 41 | 120 | 126
Suicide attempt (Psychiatric disorders) | 7 | 27 | 34
Traumatic shock (Psychiatric disorders) | 0 | 0 | 1
Voluntary hospitalization (Psychiatric disorders) | 0 | 0 | 1
Wasn't feeling well mentally (Psychiatric disorders) | 0 | 1 | 0
Separate research participation monitoring (Investigations) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 4
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4
Cold (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Flu/flu symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Lung pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 4
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 4
Rib pain/injuries (Injury, poisoning and procedural complications) | 1 | 1 | 2
Seizure (Nervous system disorders) | 3 | 8 | 6
Sexual assault/rape (Social circumstances) | 2 | 2 | 1
Shoulder injury/pain (Injury, poisoning and procedural complications) | 2 | 6 | 4
Sleep problems (General disorders) | 2 | 3 | 1
Venereal disease (Infections and infestations) | 0 | 0 | 1
stomach pain, cramps, issues, infections, ulcer (Gastrointestinal disorders) | 2 | 9 | 9
Stomach infection/flu (Infections and infestations) | 0 | 0 | 2
Fever (General disorders) | 0 | 2 | 3
Frostbite (Social circumstances) | 0 | 0 | 1
Heat exhaustion. (Social circumstances) | 0 | 1 | 0
Hypothermia (Social circumstances) | 0 | 1 | 0
Increased temperature (General disorders) | 0 | 0 | 1
Unknown medical visit (General disorders) | 3 | 11 | 9
Unknown psychiatric visit (Psychiatric disorders) | 3 | 15 | 14
Vaccinations (Surgical and medical procedures) | 0 | 1 | 1
Vehicular injury (Injury, poisoning and procedural complications) | 3 | 10 | 9
Torn ligament (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=132) | Brief Treatment (N=416) | Extended Treatment (N=408)
Ankle injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Chest pain (Cardiac disorders) | 0 | 2 | 0
Heart palpitations (Cardiac disorders) | 0 | 1 | 0
Diagnostic visits (Surgical and medical procedures) | 0 | 2 | 0
Swollen eye (Eye disorders) | 0 | 0 | 1
Fall Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal discomfort, pain, injuries (Gastrointestinal disorders) | 0 | 1 | 1
Hand injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Medication side effect: Headache (Product Issues) | 1 | 0 | 0
Medication management visit (Product Issues) | 1 | 0 | 0
Medication refilll visit (Product Issues) | 1 | 1 | 0
Lightheadness from using both NRT and cigarette use (Product Issues) | 0 | 0 | 2
NRT side effect: Discomfort (Product Issues) | 0 | 1 | 0
NRT side effect: Agitation (Product Issues) | 0 | 1 | 1
NRT side effect: Allergy to patch (Product Issues) | 0 | 0 | 2
NRT side effect: Anxiety (Product Issues) | 0 | 2 | 2
NRT side effect: Bit tongue when used nicotine gum (Product Issues) | 0 | 1 | 0
NRT side effect: Blister on tongue (Product Issues) | 0 | 1 | 0
NRT side effect: Bloating of extremities (e.g. hands, legs) (Product Issues) | 0 | 0 | 1
NRT side effect: Body ache (Product Issues) | 1 | 0 | 0
NRT side effect: Bumps on tongue (Product Issues) | 0 | 0 | 1
NRT side effect: Burning sensation (Product Issues) | 0 | 7 | 5
NRT side effect: Cold sweats (Product Issues) | 0 | 4 | 4
NRT side effect: Confusion (Product Issues) | 0 | 2 | 2
NRT side effect: Coughing (Product Issues) | 0 | 0 | 2
NRT side effect: Craving to smoke (Product Issues) | 0 | 0 | 1
NRT side effect: Diminished ability to taste (Product Issues) | 0 | 0 | 1
NRT side effect: Dizziness (Product Issues) | 2 | 15 | 13
NRT side effect: Drowsiness (Product Issues) | 0 | 1 | 0
NRT side effect: Dry mouth (Product Issues) | 1 | 2 | 5
NRT side effect: Dry skin (Product Issues) | 0 | 0 | 1
NRT side effect: Fainting (Product Issues) | 0 | 0 | 1
NRT side effect: Fatigue (Product Issues) | 1 | 1 | 0
NRT side effect: Feeling on edge (Product Issues) | 0 | 1 | 0
NRT side effect: Feeling paranoid (Product Issues) | 0 | 1 | 0
NRT side effect: Gastrointestinal distress (Product Issues) | 0 | 3 | 6
NRT side effect: Headache (Product Issues) | 1 | 14 | 16
NRT side effect: Heart burn (Product Issues) | 1 | 3 | 3
NRT side effect: Heart palpitations (Product Issues) | 0 | 8 | 8
NRT side effect: Hiccups (Product Issues) | 1 | 10 | 5
NRT side effect: Hives (Product Issues) | 0 | 1 | 0
NRT side effect: Hot flashes (Product Issues) | 0 | 1 | 0
NRT side effect: Increased appetite (Product Issues) | 0 | 0 | 2
NRT side effect: Increased saliva production (Product Issues) | 0 | 6 | 8
NRT side effect: Insomnia (Product Issues) | 1 | 12 | 11
NRT side effect: Irritability (Product Issues) | 0 | 1 | 1
NRT side effect: Irritation on body (Product Issues) | 0 | 1 | 2
NRT side effect: Itchiness (Product Issues) | 7 | 32 | 29
NRT side effect: Jaw muscle aches (Product Issues) | 2 | 3 | 1
NRT side effect: Jaw tightness (Product Issues) | 0 | 0 | 1
NRT side effect: Jitteriness (Product Issues) | 0 | 1 | 2
NRT side effect: Lightheadedness (Product Issues) | 0 | 11 | 7
NRT side effect: Localized pain where patch was (Product Issues) | 0 | 1 | 0
NRT side effect: Migraines (Product Issues) | 0 | 1 | 0
NRT side effect: Mild buzz (Product Issues) | 0 | 0 | 1
NRT side effect: More prone to migraines (Product Issues) | 0 | 0 | 1
NRT side effect: Mouth sores (Product Issues) | 1 | 2 | 1
NRT side effects: Muscle cramps (Product Issues) | 0 | 1 | 0
NRT side effect: Nausea (Product Issues) | 3 | 31 | 22
NRT side effect: Nervousness (Product Issues) | 0 | 2 | 0
NRT side effect: Nicotine rush and crash (Product Issues) | 0 | 0 | 1
NRT side effect: Nightmares (Product Issues) | 0 | 3 | 1
NRT side effects: Numbness (Product Issues) | 0 | 1 | 1
NRT side effect: Peppery burning (Product Issues) | 0 | 0 | 1
NRT side effect: Perspiration (Product Issues) | 0 | 1 | 3
NRT side effect: Rash (Product Issues) | 0 | 2 | 2
NRT side effect: Red circle on skin (Product Issues) | 0 | 1 | 0
NRT side effect: Red tiny blisters when patch was applied to sensitive skin (i.e. under arm) (Product Issues) | 0 | 1 | 0
NRT side effect: Redness (Product Issues) | 4 | 20 | 12
NRT side effect: Sharp joint pain (Product Issues) | 0 | 1 | 0
NRT side effect: Shortness of breath (Product Issues) | 0 | 0 | 1
NRT side effect: Skin irritation (Product Issues) | 2 | 0 | 4
NRT side effect: Soreness (Product Issues) | 0 | 0 | 1
NRT side effect: Sticky Residue (Product Issues) | 1 | 0 | 0
NRT side effect: Stinging sensation (Product Issues) | 0 | 0 | 2
NRT side effect: Stomachache (Product Issues) | 3 | 13 | 2
NRT side effect: Swelling (Product Issues) | 0 | 3 | 4
NRT side effect: Throat irritation (Product Issues) | 0 | 1 | 3
NRT side effect: Trouble urinating (Product Issues) | 0 | 0 | 1
NRT side effect: Uncomfortable stimulation (Product Issues) | 0 | 0 | 1
NRT side effect: Vivid dreams/nightmares (Product Issues) | 2 | 21 | 23
NRT side effect: Vomiting (Product Issues) | 0 | 3 | 5
NRT side effect: Watery stool (Product Issues) | 0 | 1 | 0
NRT side effect: Weird dreams (Product Issues) | 0 | 2 | 1
Occupational injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Abdominal discomfort (General disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diabetes (Metabolism and nutrition disorders) | 0 | 0 | 1
Diarrhea (Renal and urinary disorders) | 0 | 1 | 0
Excessive vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Symptoms of hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0
Hemorrhoids (Renal and urinary disorders) | 1 | 0 | 0
Migraines (General disorders) | 0 | 1 | 0
Muscle aches (General disorders) | 0 | 1 | 0
Shingles (Infections and infestations) | 1 | 0 | 0
Unable to eat (General disorders) | 0 | 1 | 0
Psychiatric evaluation (Social circumstances) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Issues with housing staff (Social circumstances) | 0 | 0 | 1
Mood lability, disorganized behavior (Psychiatric disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Confusion/Disorientation (Psychiatric disorders) | 0 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Broken ribs (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Substance use related events (Psychiatric disorders) | 1 | 1 | 2
Surgery (Surgical and medical procedures) | 0 | 0 | 1
Vehicular injury (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No